CLINICAL TRIAL: NCT04718038
Title: A Clinical Study of Continuing Cetuximab Plus Chemotherapy After First Progression in Wild-type KRAS, NRAS and BRAF V600E Metastatic Colorectal Cancer
Brief Title: Continuing Cetuximab Plus Chemotherapy After First Progression in Wild-type KRAS, NRAS and BRAF V600E Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HNCH-GI-100
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Wild-type KRAS,NRAS and BRAF V600E Metastatic Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cetuximab combind mFOLFOX6/FOLFIRI — Cetuximab 500mg/m2 ivgtt 2h d1 ,q14d;mFOLFOX6: Oxaliplatin 85mg/m2 ivgtt 2h d1, 5-Fu 400mg/m2 iv d1,Lefucovorin 400mg/m2 ivgtt 2h d1, 5-Fu 2.4/m2 CIV 46h, q14d; FOLFIRI: CPT-11 180mg/m2 ivgtt 60-90mins d1, 5-Fu 400mg/m2 iv d1,Lefucovorin 400mg/m2 ivgtt 2h d1,5-Fu 2.4/m2 CIV 46-48h, q14d

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of continuing cetuximab combined with chemotherapy after first-line progression in wild-type KRAS,NRAS and BRAF colorectal cancer.

DETAILED DESCRIPTION:
In addition to the sequential therapeutic schedule of offering maintenance therapy and reintroduction of chemotherapy regimens to patients with nonresectable mCRC, multiline treatment strategy of continuing bevacizumab after progression to first-line bevacizumab plus chemotherapy demonstrated optimal clinical benefits in prolonging progression-free survival (PFS) and overall survival (OS) . Continuing cetuximab after progression to first-line cetuximab is also a promising strategy. The underlying hypothesis is that a sustained inhibition of EGFR signaling with cetuximab would continuously eliminate sensitive clones of RAS wild-type tumor. The present phase 2 clinical trial evaluated standard fluoropyrimidine-based chemotherapy combined with cetuximab among patients with wild-type KRAS, NRAS and BRAF V600E mCRC who had progressed after cetuximab plus standard chemotherapy in the first-line setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent.
2. Patients with wild-type KRAS,NRAS and BRAF V600E metastatic colorectal adenocarcinoma confirmed by histology and genetic testing.
3. Patients with metastatic colorectal cancer (stage IV) confirmed by imaging (CT/MRI) with measurable lesions (according to RECIST 1.1 criteria)
4. Patients who had previously received first-line standard chemotherapy in combination with cetuximab, or/and maintenance therapy with cetuximab for disease progression.The standard treatment regimens include XELOX, FOLFOX, and FOLFIRI.

5.18-70 years old ;ECOG PS score: 0~1;Life expectancy ≥ 12 weeks. 6. Provide histological specimens for secondary detection: primary lesion or metastatic lesion.

7.The main organ function meets the following criteria within 7 days before treatment:

(1)Blood routine examination criteria (without blood transfusion within 14 days): Hemoglobin (HB) ≥ 90g / L; The absolute value of neutrophils (ANC) ≥ 1.5 × 109 / L; Platelet (PLT) ≥ 80 × 109 / L; (2) Biochemical examinations must meet the following criteria: Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) ≤ 2.5 * ULN; serum creatinine (Cr) ≤ 1.5 * ULN or creatinine clearance (CCr) ≥ 60ml / min; (3) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).

8.Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating patients; men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1. Exceeding or currently suffering from other malignant tumors within 5 years, except for cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (in situ carcinoma) And T1 (tumor infiltrating basement membrane)].
2. Radiation therapy on tumor target was performed within 4 weeks before enrollment.
3. Unmitigated toxic reactions higher than CTC AE(4.0) grade 2 or above due to any prior treatment, excluding alopecia and neurotoxicity ≤ grade 2 due to oxaliplatin.
4. Any severe and/or uncontrolled disease, including:

   1. patients with hypertension who are not well controlled by antihypertensive drug (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg).
   2. with grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification).
   3. Severe or uncontrolled disease or active infection (≥CTCAE grade 2 infection), which the investigator believes may increase the risk associated with study participation, study drug administration, or affect the subject's ability to receive study medication.
   4. Renal failure requires hemodialysis or peritoneal dialysis.
   5. a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
   6. Patients with diabetes who have poor glycemic control (fasting blood glucose (FBG) > 10 mmol/L); subjects with active, known or suspected autoimmune diseases. Subjects with type 1 diabetes, residual hypothyroidism caused by autoimmune thyroiditis requiring hormone replacement therapy, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia) can be enrolled.
   7. patients with seizures and requiring treatment.
5. Patients with gastrointestinal diseases such as intestinal obstruction (including incomplete intestinal obstruction) or those who may have caused gastrointestinal bleeding, perforation or obstruction.
6. Patients who underwent surgical treatment, incisional biopsy or significant traumatic injury within 28 days prior to enrollment.
7. In the 4 weeks prior to enrollment, patients with any bleeding event ≥ CTCAE 3 have unhealed wounds, ulcers or fractures.
8. Overactive/venous thrombosis events within 3 months, such as cerebrovascular accidents (including transient ischemic attacks), deep static Pulmonary thrombosis and pulmonary embolism.
9. those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder.
10. Patients with brain metastases.
11. Patients who have participated in other clinical trials of anti-tumor drugs within four weeks.
12. According to the investigator's judgment, there is a concomitant disease that seriously harms the patient's safety or affects the patient's completion of the study.
13. Cannot perform biopsy to provide histological specimens.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2020-09-01

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  The time from randomization to documented disease progression or death from any cause

SECONDARY OUTCOMES:
Overall Survial(OS) | 2 years
  The time from randomization to death from any cause
ORR | 2 years
  The percentage of complete or partial responses
Safety | 2 years
  assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events [version 3.0]